CLINICAL TRIAL: NCT03754543
Title: Iron Bioavailability From Fortified Cereal in Malawian Infants
Brief Title: Baby Iron Bioavailability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Swiss Federal Institute of Technology (Other); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 18.05.INF
Record Dates: First submitted 2018-10-04; First posted 2018-11-27 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Iron Bioavailability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Testmeal A (Active Comparator): A new, whole-grain infant cereal fortified with ferrous fumarate
  Interventions: Other: Labeled iron salt Fe54
- Testmeal B (Active Comparator): An alternative new whole-grain infant cereal recipe fortified with ferrous fumarate
  Interventions: Other: Labeled iron salt Fe57
- Testmeal C (Placebo Comparator): An existing, refined grain infant cereal fortified with ferrous fumarate
  Interventions: Other: Labeled iron salt Fe54
- Testmeal D (Active Comparator): An existing, whole-grain infant cereal fortified with ferrous fumarate
  Interventions: Other: Labeled iron salt Fe57
- Testmeal E (Active Comparator): An existing, whole-grain infant cereal fortified with ferrous bisglycinate
  Interventions: Other: Labeled iron salt Fe58

INTERVENTIONS:
Other: Labeled iron salt Fe54 — Ferrous fumarate enriched with Fe 54 isotopes contains 2.25 mg of iron source and 13.5 mg of Vitamin C per serving
  Arms: Testmeal A; Testmeal C
Other: Labeled iron salt Fe57 — Ferrous fumarate enriched with Fe 57 isotopes contains 2.25 mg of iron source and 13.5 mg of Vitamin C per serving
  Arms: Testmeal B; Testmeal D
Other: Labeled iron salt Fe58 — Ferrous bisglycinate enriched with Fe 58 isotopes contains 2.25 mg of iron source and 13.5 mg of Vitamin C per serving
  Arms: Testmeal E

SUMMARY:
The overall objective of this trial is to investigate the iron bioavailability from new infant cereals in Malawian infants.

DETAILED DESCRIPTION:
In 30 infants aged 6 to 14 months old, the investigator will administer in random order over 2 phases separated by 14 days, 5 infant cereals containing either ferrous fumarate (4 meals) or ferrous bisglycinate (1 meal) intrinsically labeled with stable isotopes. The investigator will collect one blood sample at baseline and another sample at the end of each phase, thus 3 samples total. In these samples, fractional iron absorption and markers of iron and inflammation status will be measured . In addition, infant and child acceptability of one of the infant cereals will be assessed by using a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Infant age 6 - 14 months
2. Infant exhibits no clinical signs / symptoms of chronic disease or acute illness
3. Capillary haemoglobin concentration > 70g/L
4. Z-scores for weight-for-age and weight-for-length > -2
5. Infant's parent(s) / legally acceptable representative is of legal age of consent, has anticipated residence in the area for the duration of the study, and is willing and able to fulfil the requirements of the study protocol
6. Infant is expected to consume the entire 25 g portion during infant cereal feeding based on the Investigator's judgement established via observations of feeding during the adaptation phase
7. Infant received a complete dose of intermittent preventive treatment with dihydroartemisinin piperaquine (IPTi-DP) as well a single dose of antihelminth treatment with Albendazole

Exclusion Criteria:

1. Parents not willing / not able to comply with the requirements of study protocol
2. Infants receiving iron-containing supplements in the 2 months prior to enrollment (other supplements are acceptable)
3. Infants with allergies or intolerance to wheat, oat, gluten or other ingredients in the test cereals (e.g., celiac disease)
4. Infants participating in any other clinical trial prior to enrollment
5. Infants or infant's family who in the Investigator's judgment cannot be expected to comply with the protocol or study procedures.

Ages: 6 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption of 54FeFum (test cereal A), 57FeFum (test cereal B), 54FeFum (test cereal C). | up to 6 weeks
  Fractional iron absorption of 54FeFum (test cereal A), 57FeFum (test cereal B), 54FeFum (test cereal C). Based on the shift of Fe isotope ratios in the blood samples and the amount of Fe circulating in the body, the amounts of 54Fe and 57Fe isotopic label present in the blood 14 days after the test meal administrations will be calculated on the principle of isotope dilution and considering that the iron isotopic labels are not mono-isotopic

SECONDARY OUTCOMES:
Fractional iron absorption of 54FeFum (test cereal C), 57FeFum (test cereal D), 58FeBisGly (test cereal E). | up to 6 weeks
  Fractional iron absorption of 54FeFum (test cereal C), 57FeFum (test cereal D), 58FeBisGly (test cereal E). Based on the shift of Fe isotope ratios in the blood samples and the amount of Fe circulating in the body, the amounts of 54Fe, 57Fe and 58Fe isotopic label present in the blood 14 days after the test meal administrations will be calculated as described above for the primary endpoint
Cereal acceptability questionnaire | up to 2 weeks
Fractional iron absorption from infants with (CRP ≥ 10 mg/L) or without (CRP < 10 mg/L) asymptomatic infection / inflammation. | up to 6 weeks
Standard reporting of adverse events (AEs) for safety assessment | time of consent to 24 hours after final blood draw
  Reported AEs will include type, incidence, severity, seriousness and relation to intervention. All concomitant medications used to treat illnesses and other conditions will be recorded (both dose and duration).

CONTACTS AND LOCATIONS:
Overall Officials: Kamija Phiri, Prof., Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- Central Hospital, Zomba, Malawi

IPD SHARING:
Plan to Share IPD: No